CLINICAL TRIAL: NCT02103348
Title: Characterizing Asthma Sputum Elasticity in the UCSF Severe Asthma Research Program
Acronym: CAESAR
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 14-13242
Record Dates: First submitted 2014-03-24; First posted 2014-04-03 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: Severe asthma; Sputum; Mucolysis
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of induced sputum and blood for DNA and RNA extraction, plasma, and serum will be banked in the UCSF Airway Tissue Bank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild-to-Moderate Asthma: Those with mild-to-moderate persistent asthma as defined by the NAEPP EPR-3 guidelines.
- Severe Asthma: Major Criteria: (1 required)
  1. Treatment with oral corticosteroids for at least 6 of the previous 12 months
  2. Treatment with high-dose inhaled corticosteroids for at least 10 of the previous 12 months
  Minor Criteria: (2 required)
  1. Daily treatment with an asthma controller medication in addition to inhaled, or
  2. Asthma symptoms requiring short-acting bronchodilator use on a daily or near daily basis (defined as at least 5 of 7 days), or
  3. Persistent airway obstruction with baseline FEV1 <80% predicted, or
  4. ≥ 1 urgent visits for asthma in the previous 12 months, or
  5. ≥ 3 systemic corticosteroid bursts in the previous 12 months, or
  6. Prompt deterioration with a reduction in oral or inhaled corticosteroid dose, or
  7. A near-fatal asthma event (i.e., intubation) in the past.
- Healthy Controls: Those without asthma or other chronic lung disease.

SUMMARY:
This study is designed to characterize subjects in terms of their sputum phenotype. The purpose of this study is to learn more about the impact of having abnormally elastic sputum on asthma severity by comparing subjects with severe as well as mild/moderate asthma to healthy controls. The characterization will include medical history, pulmonary function testing, imaging of the lungs and biospecimen collection.

DETAILED DESCRIPTION:
Asthma is a heterogeneous disease characterized by airway hyperreactivity and chronic airway inflammation. Published literature from the last few years has shown that asthma does not behave like a single disease but is more of a syndrome with vast heterogeneity in pathogenesis, severity, and treatment response. Various clinical phenotypes and endotypes have been described that advance our understanding of these differences and the mechanisms underlying them. We propose there is a subgroup of asthmatic patients that have sputum with abnormal biophysical properties. Healthy airway mucus is composed of a lightly cross-linked gel that is easily transported by the mucociliary apparatus, coughed and expectorated or swallowed. Pathologic mucus has, in contrast, abnormally high elasticity. This is due to a more cross linked structure which gives the sputum the properties of solid and makes sputum difficult to mobilize. Increased sputum elasticity makes expectoration of sputum more difficult and leads to airflow obstruction. Pathologic mucus contributes to airflow obstruction and airway infection in multiple lung diseases, including asthma. Mucus plugs are a particular problem in asthmatic patients with allergic bronchopulmonary aspergillosis (ABPA)The identification of phenotype of severe asthma with pathologic mucus contributing to disease severity may change how we think about severe asthma, moving towards therapies targeting mucus clearance such as in other conditions such as cystic fibrosis. Pathologic mucus in severe asthma is characterized by cellular inflammation, high concentrations of mucins and DNA polymers. Knowledge of specific cellular and biochemical constituents of pathologic mucus in severe asthma can guide targeted mucolytic treatment with n-acetylcysteine, rhDNAse, or novel mucolytic agents.

As part of the Severe Asthma Research Program (SARP), UCSF is in a unique position to recruit a large number of severe asthmatic subjects within which we expect a portion will demonstrate high sputum elasticity. We will also through CAESAR recruit additional subjects with moderate to severe airflow obstruction. We will perform rheological measurement on all subjects that are recruited to our site and from this identify a group of asthmatic cases that have an elastic modulus of ≥1 or <1 and compare properties of sputum from these subjects to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 bronchodilator reversibility ≥12% or airway hyperresponsiveness reflected by a methacholine PC20 ≤16 mg/mL
* An exception will be made for enrollees whose FEV1 is < 50% predicted (<70% in children aged 6 to 17 years), precluding methacholine challenge testing. If bronchodilator reversibility is <12% in these participants, a diagnosis of asthma acceptable to the investigator is sufficient for inclusion in CAESAR.

Exclusion Criteria:

* Pregnancy,
* Current smoking,
* Smoking history > 10 pack years if ≥30 years of age, or smoking history > 5 pack years if <30 years of age,
* Other chronic pulmonary disorders associated with asthma-like symptoms, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction (that is the sole cause of respiratory symptoms and at the PI's discretion), severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways,
* History of premature birth before 35 weeks gestation,
* Planning to relocate from the clinical center area before study completion,
* Any other criteria that place the subject at unnecessary risk according to the judgment of the Principal Investigator and/or attending physician(s) of record, or
* Currently participating in an investigational drug trial.

Healthy Controls:

Inclusion criteria: Healthy subjects between the age of 18y and 65y. At least 3 of the 7 subjects per center should be aged 35y or older.

Exclusion criteria

* History of chronic diseases that affect the lungs.
* A history suggestive of allergic rhinitis, eczema or chronic sinusitis.
* An improvement in FEV1 of more than 12% following 4 puffs of albuterol.
* Smoking history > 10 pack years if ≥30 years of age, or smoking history > 5 pack years if <30 years of age, or any smoking within the past year.
* Respiratory tract infection within the past 4 weeks.
* Pregnancy.
* History of premature birth (<35 weeks).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A diverse sample of subjects with asthma is needed to gain better understanding of asthma and its endotypes. CAESAR will therefore enroll subjects between 18 and 65 years with a physician diagnosis of asthma as well as a group of healthy subjects. The target recruitment goal for UCSF is 50 adults with asthma and 25 healthy controls (age 18 and older). Within the asthma group, an attempt will be made to enroll 60% of subjects with severe with the rest of the subjects mild to moderate asthma.Within the cohort, an attempt will be made to enroll at least 50% females and 10% minorities.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Lung function | Cross sectional over 4-6 weeks
  Lung function as a measure of asthma severity.

SECONDARY OUTCOMES:
Inflammatory cellular markers | Cross sectional over 4-6 weeks
  Changes in inflammatory cellular markers in sputum and blood. We will measure various indicators of airway inflammation and compare them with various phenotypic characteristics.

OTHER OUTCOMES:
CT Chest | Cross sectional over 4-6 weeks
  Examining CT chest in asthmatics for evidence of retained mucus.

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, M.D. M.SC., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: Airway Clinical Research Center website — http://acrc.ucsf.edu